CLINICAL TRIAL: NCT01172223
Title: Phase I/II Trial of Primary Chemotherapy With Non-pegylated Liposomal Doxorubicin, Paclitaxel and Lapatinib in Patients With HER2-positive Early
Brief Title: Primary Chemotherapy in Patients With HER2-positive Early Breast Cancer
Acronym: LAPADO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof Dirk Elling (Other)
Responsible Party: Sponsor-Investigator, Prof Dirk Elling, Professor, Sana-Klinikum Lichtenberg
Organization: Sana-Klinikum Lichtenberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAPADO-Study; 2007-000924-42 (EudraCT Number)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: HER2-positive; early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Paclitaxel; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAPADO (Experimental): Non-pegylated liposomal doxorubicin (NPLD; Myocet, 60 mg/m2 i.v. day 1 q3 weeks), Paclitaxel (175 mg/m2 i.v. day 1 q3 weeks), and Lapatinib (GW572016, Tykerb, 750-1500 mg/d orally daily until the day of the definitive surgery)
  Interventions: Drug: Myocet (Non-pegylated liposomal doxorubicin (NPLD)); Drug: Paclitaxel; Drug: Lapatinib (GW572016, Tykerb)

INTERVENTIONS:
Drug: Myocet (Non-pegylated liposomal doxorubicin (NPLD)) — 60 mg/m^2 i.v. day 1 q3 weeks
Drug: Paclitaxel — 175 mg/m^2 i.v. day 1 q3 weeks
Drug: Lapatinib (GW572016, Tykerb) — 750-1500 mg/d orally daily until the day of the definitive surgery

SUMMARY:
Open-label, multicenter phase I/II trial. Patients with HER2-positive (overexpressing or amplified), invasive breast cancer with T1c N1-2 or T2 N0-2 disease will be treated with

* Non-pegylated liposomal doxorubicin (NPLD; Myocet, 60 mg/m^2 i.v. day 1 q3 weeks),
* Paclitaxel (175 mg/m^2 i.v. day 1 q3 weeks), and
* Lapatinib (GW572016, Tykerb, 750-1500 mg/d orally daily until the day of the definitive surgery) Treatment is planned for 6 cycles unless there is evidence of unacceptable toxicity, disease progression or inadequate efficacy (defined as a decrease in tumor size <25% after 4 courses measured by ultrasound or MR-mammography), or if the patient requested to be released.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy affecting females in northern Europe and North America, corresponding to an age-corrected annual incidence of 100 to 120 per 100000 females. Approximately 30-40% of all patients treated with curative intent will develop metastatic disease. Perioperative systemic treatment has made a major impact on relapse-free and overall survival of women with early-stage breast cancer [ , ] with therapeutic strategies being based on the endocrine responsiveness and the estimated risk of relapse defined by tumor size, axillary lymph node involvement, histologic and nuclear grade, lymphatic and/or vascular invasion, HER2/neu-overexpression and age [ ]. Perioperative therapy has traditionally been administered postoperatively, but chemotherapy is increasingly utilized in the preoperative setting as it can significantly improve the rate of breast conserving surgery, and new regimens can be evaluated rapidly and more precisely.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* T1c N1-2 or T2 N0-2 disease
* HER2-positive tumours with 3+ intensity on immunohistochemical staining for HER2 or amplification of the HER2 gene on fluorescence in situ hybridization (FISH)
* No prior systemic treatment regimens for breast cancer
* Adequate hematologic function (ANC 1500 cells/µl, platelet count 100000/µl, and hemoglobin 8g/dl).
* Serum creatinine concentration < 1.5 times the upper limit of normal (ULN) and/or creatinine clearance >60 ml/min
* Bilirubin level < 1.5 X ULN
* Normal cardiac function with a left ventricular ejection fraction of at least 50% (as assessed by quantitative echocardiogram or MUGA scan)
* Karnofsky performance status 80%
* Age 18 years
* If the patient is of childbearing potential, she agrees to: comply with effective contraceptive measures, has been using adequate contraception since the last menses, will use adequate contraception during the study, and has a negative pregnancy test within one week of study entry
* Written informed consent prior to admission to this study

Exclusion Criteria:

* Male patients
* Inflammatory or bilateral breast cancer
* Evidence of distant metastases
* Previous systemic or local treatment for breast cancer (including surgery, radiotherapy, cytotoxic and endocrine treatments)
* Past or current history of other neoplasms, except for
* Curatively treated non-melanoma skin cancer
* Adequately treated in situ carcinoma of the cervix
* Other cancer curatively treated and with no evidence of disease for at least 5 years
* Significant cardiac disease, including angina pectoris, severe cardiac arrhythmia requiring medication, severe conduction abnormalities, clinically significant valvular disease, cardiomegaly, ventricular hypertrophy, poorly uncontrolled hypertension (resting diastolic blood pressure >115 mmHg), prior myocardial infarction, CHF, or other cardiomyopathy
* Preexisting sensoric or motor polyneuropathy Grade 2 according to NCI CTC
* Serious intercurrent medical or psychiatric illness, including serious active infection
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study entry.
* Detained persons or prisoners
* Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Determine the optimal doses for NPLD, paclitaxel and lapatinib (phase I) | every 3 weeks
Evaluate the pathological response to NPLD, paclitaxel and lapatinib (phase II) | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elling, Principal Investigator — Sana Klinikum Lichtenberg, Berlin
Locations (1):
- Sana Klinikum Lichtenberg, Berlin, Germany